CLINICAL TRIAL: NCT06972758
Title: A Phase II Study of EVEerolimus as Adjuvant Therapy After Surgical Resection for Hepatocellular cArcinoma at High Risk of RecurreNCE [SEVERANCE Trial]
Brief Title: Adjuvant Everolimus in High-Risk Hepatocellular Carcinoma After Curative Resection (SEVERANCE Trial)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2025-0275
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Carcinom; Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treamtent group (Experimental): Patients recieving study drug
  Interventions: Drug: Certirobell®

INTERVENTIONS:
Drug: Certirobell® — Patients enrolled in the study will initiate oral administration of Certirobell® between 4 to 6 weeks after hepatic resection. The medication will be taken for a duration of 92 weeks, twice daily at approximately 12-hour intervals. The initial dosage is 1.0 mg per dose (twice daily). For patients with a Child-Pugh score of 6, the starting dose will be reduced to 0.75 mg per dose (twice daily). At each visit, the blood concentration of Certirovel will be measured, and the investigator will adjust the dosage as needed to maintain levels within the target range of 3-8 ng/mL. If HCC recurrence is confirmed during treatment, the administration of the drug will be discontinued.

SUMMARY:
"Hepatic resection is the primary curative treatment for patients with a single, liver-confined hepatocellular carcinoma (HCC) without cirrhosis and is also considered in patients with cirrhosis if residual liver function is sufficient. Despite curative resection, HCC has a high recurrence rate, with 5-year recurrence reported in approximately 50-70% of patients. Notably, in cases with microvascular invasion, the 2-year recurrence rate reaches 55-75%. As early recurrence strongly impacts overall survival, there is a critical need for effective adjuvant therapies; however, no adjuvant treatment has yet been established or officially recommended.

Everolimus is an mTOR inhibitor that has both immunosuppressive and antitumor effects. Approximately half of HCC cases exhibit activation of the mTOR pathway. In liver transplant recipients, everolimus is used as an immunosuppressive agent and has been associated with reduced recurrence and improved survival, particularly in patients with elevated tumor markers prior to transplantation. Preclinical studies at our institution have shown that mTOR inhibitors may be more effective in preventing tumor development than in treating established tumors, suggesting a potential benefit for everolimus in an adjuvant setting.

To date, no clinical trials have assessed the efficacy of everolimus as adjuvant therapy after curative hepatic resection, especially in high-risk HCC characterized by microvascular invasion or satellite nodules. This study aims to evaluate the efficacy and safety of everolimus (Certirobell®) as adjuvant therapy in high-risk HCC patients following curative resection.

This is a single-center, single-arm Phase II trial conducted at Severance Hospital. A total of 60 patients with pathologically confirmed HCC who underwent R0 resection and exhibit high-risk features for recurrence will be enrolled. Everolimus will be administered orally, twice daily for 92 weeks, starting 4 to 6 weeks postoperatively. Initial dosing will be 1.0 mg twice daily, adjusted to 0.75 mg for patients with a Child-Pugh score of 6. Dosage adjustments will be made based on everolimus trough levels, targeting 3-8 ng/mL. Treatment will be discontinued upon confirmation of HCC recurrence.

The primary endpoint is 2-year recurrence-free survival (RFS). Secondary endpoints include 1-year RFS, 2-year recurrence rate, overall survival (OS), time to recurrence, and safety outcomes.

An interim analysis will be conducted after the first 30 patients have been enrolled and followed for 2 years. Based on the interim assessment of efficacy or futility, the study will either be terminated early or proceed with enrollment of an additional 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Alkaline phosphatase level > 2.5 times the ULN
* Proteinuria defined as a urine protein-to-creatinine ratio > 1.0 g/gCr or ≥ 2+ on urine dipstick
* Patients who received systemic therapy prior to hepatic resection
* Prior treatment with anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapies
* Renal impairment with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m² (based on MDRD formula)
* Total cholesterol > 350 mg/dL or triglycerides > 500 mg/dL
* History of severe acute (within the past 4 weeks) or chronic hypersensitivity reactions requiring treatment to everolimus or drugs with a similar chemical structure
* Pregnant or breastfeeding women, women who are possibly pregnant, or women of childbearing potential who are unable to use highly effective contraception† during the study period and for 8 weeks after the last dose
* Any condition deemed by the investigator to render the patient unsuitable for participation in the clinical trial

  * Highly effective contraception is defined as methods with a failure rate of less than 1% per year, including bilateral tubal occlusion, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUDs), and copper IUDs. Methods such as calendar-based methods, ovulation prediction, symptothermal methods, and post-ovulation methods are not considered adequate contraception.

Exclusion Criteria:

* Patients diagnosed with combined hepatocellular-cholangiocarcinoma (HCC-CCC)
* Presence of clinically significant ascites
* History of hepatic encephalopathy
* History of variceal bleeding within 6 months prior to hepatic resection
* Autoimmune diseases or immunodeficiency disorders
* Serious cardiovascular diseases, including acute myocardial infarction, acute coronary syndrome, stroke, or heart failure of New York Heart Association (NYHA) Class II or higher
* History of malignancies other than HCC within the past 5 years
* Patients with hereditary metabolic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Patients currently taking medication for psychiatric disorders
* Absolute neutrophil count (ANC) < 1500/μL or platelet count < 75,000/μL
* AST, ALT, or total bilirubin levels > 3 times the upper limit of normal (ULN)
* Alkaline phosphatase level > 2.5 times the ULN
* Proteinuria defined as a urine protein-to-creatinine ratio > 1.0 g/gCr or ≥ 2+ on urine dipstick
* Patients who received systemic therapy prior to hepatic resection
* Prior treatment with anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapies
* Renal impairment with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m² (based on MDRD formula)
* Total cholesterol > 350 mg/dL or triglycerides > 500 mg/dL
* History of severe acute (within the past 4 weeks) or chronic hypersensitivity reactions requiring treatment to everolimus or drugs with a similar chemical structure
* Pregnant or breastfeeding women, women who are possibly pregnant, or women of childbearing potential who are unable to use highly effective contraception† during the study period and for 8 weeks after the last dose
* Any condition deemed by the investigator to render the patient unsuitable for participation in the clinical trial

  * Highly effective contraception is defined as methods with a failure rate of less than 1% per year, including bilateral tubal occlusion, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUDs), and copper IUDs. Methods such as calendar-based methods, ovulation prediction, symptothermal methods, and post-ovulation methods are not considered adequate contraception.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | 2-year from hepatic resection
  The 2-year recurrence-free survival (RFS) is defined as the proportion of patients who remain alive without intrahepatic or extrahepatic recurrence at 2 years from the time of hepatic resection.

IPD SHARING:
Plan to Share IPD: No